CLINICAL TRIAL: NCT01815281
Title: Foot Mechanical Stimulation for Treatment of Gait and Gait Related Disorders in Parkinson's Disease
Brief Title: Foot Mechanical Stimulation for Treatment of Gait and Gait Related Disorders in Parkinson's Disease and Progressive Supranuclear Palsy.
Acronym: GONDOLAPILOTA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele Roma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RP 12/13
Record Dates: First submitted 2013-03-14; First posted 2013-03-21 (Estimated); Last update posted 2024-04-10 (Actual); Status verified 2015-03

CONDITIONS: Idiopathic Parkinson's Disease; Progressive Supranuclear Palsy
MeSH Terms: conditions — Parkinson Disease; Supranuclear Palsy, Progressive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Foot Mechanical Stimulation (Experimental): The FMS stimulation will be given to all participants using GONDOLA equipment (Ecker Technologies Sagl, Switzerland).
  Interventions: Device: Foot Mechanical Stimulation (GONDOLA)
- Footh Mechanical Stimulation (Sham Comparator): The sham stimulation will be given to all participants using GONDOLA equipment (Ecker Technologies Sagl, Switzerland).
  Interventions: Device: Foot Mechanical Stimulation (GONDOLA)

INTERVENTIONS:
Device: Foot Mechanical Stimulation (GONDOLA)
  Other Names: GONDOLA equipment (Ecker Technologies Sagl, Switzerland).

SUMMARY:
The purpose of this research study is to evaluate safety and effectiveness of Foot Mechanical stimulation to improving Gait and Gait Related Disorders in Parkinson Disease and Progressive Supranuclear Palsy both stable and with motor fluctuation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic PD or PSP by UK Brain Bank criteria,
* Able to walk 25 feet unassisted or with minimal assistance;
* On stable doses of Parkinson's medications for at least 2 weeks prior to study onset;
* Endurance sufficient to stand at least 20 minutes unassisted per patient report.

Exclusion Criteria:

* Other significant neurological or orthopedic problems.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-07; Primary Completion 2013-11 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go. | Change from Baseline in Timed Up and Go test at 1 month follow up.
  Time Up and Go test will be collected in OFF state 4 hour after oral assumption of levodopa at baseline (inclusion) (T0), before (T1-T3-T5-T7-T9-T11) and after all stimulation (T2-T4-T6-T8-T10) and endpoint (after 6 stimulation) (T12) at the follow-up examination after 1 months from the treatments conclusion (T13).

SECONDARY OUTCOMES:
6 minuts walking test. | Change from Baseline in gait speed at 1 month follow up
  6 minuts walking test will be collected in OFF state 4 hour after oral assumption of levodopa at baseline (inclusion) (T0), before (T1-T3-T5-T7-T9-T11) and after all stimulation (T2-T4-T6-T8-T10) and endpoint (after 6 stimulation) (T12) at the follow-up examination after 1 months from the treatments conclusion (T13).
Gait Parameters | Change from Baseline in Gait Parameters at 1 month follow up
  Gait Analysis will be collected in OFF state 4 hour after oral assumption of levodopa at baseline (inclusion) (T0), before (T1-T3-T5-T7-T9-T11) and after all stimulation (T2-T4-T6-T8-T10) and endpoint (after 6 stimulation) (T12) at the follow-up examination after 1 months from the treatments conclusion (T13).
FREEZING OF GAIT QUESTIONNAIRES | Change from Baseline in FREEZING OF GAIT QUESTIONNAIRES at 1 month follow up.
THE PARKINSON'S DISEASE QUESTIONNAIRE (PDQ-39) | Change from Baseline in PDQ-39 at 1 month follow up

OTHER OUTCOMES:
UNIFIED PARKINSON'S DISEASE RATING SCALE (UPDRS). | Change from Baseline in UPDRS scores at 1 month follow up
PROGRESSIVE SUPRANUCLEAR PALSY RATING SCALE (PSP RATING SCALES) | Change from Baseline in PSP RATING SCALES scores at 1 month follow up
Functional Ambulation classification (FAC) | Change from Baseline in FAC scores at 1 month follow up
Walking handicap Scale (WHS) | Change from Baseline in WHS scores at 1 month follow up
BOLD signal response to gondola treatment | Change from Baseline in UPDRS scores at 1 month follow up
  BOLD signal will be collected in OFF state 4 hour after oral assumption of levodopa at baseline (inclusion) (T0), before (T1-T3-T5-T7-T9-T11) and after all stimulation (T2-T4-T6-T8-T10) and endpoint (after 6 stimulation) (T12) at the follow-up examination after 1 months from the treatments conclusion (T13).

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio Stocchi, MD, Principal Investigator — IRCCS San Raffaele Pisana Rome Italy; Michela Goffredo, BME, Study Director — IRCCS San Raffaele Pisana Rome Italy
Locations (3):
- Italy (3):
  - San Raffaele Cassino, Cassino, FR
  - University Campus Biomedico of Rome, Rome
  - IRCCS San Raffaele Roma, Rome

REFERENCES:
- [Derived] Quattrocchi CC, de Pandis MF, Piervincenzi C, Galli M, Melgari JM, Salomone G, Sale P, Mallio CA, Carducci F, Stocchi F. Acute Modulation of Brain Connectivity in Parkinson Disease after Automatic Mechanical Peripheral Stimulation: A Pilot Study. PLoS One. 2015 Oct 15;10(10):e0137977. doi: 10.1371/journal.pone.0137977. eCollection 2015. PMID 26469868